CLINICAL TRIAL: NCT06447961
Title: The Psychological Impacts of Living With an Inherited Colorectal Cancer Predisposition Syndrome
Brief Title: PSYLIVED: the Psychological Impacts of Living With an Inherited Colorectal Cancer Predisposition Syndrome
Acronym: PSYLIVED
Status: Recruiting | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RD23/130; 326731 (Other: IRAS)
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Lynch Syndrome; Polyposis Syndrome, Hereditary Mixed, 1; Polyposis Syndrome, Hereditary Mixed, 2
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Polyposis Syndrome, Hereditary Mixed, 1; Polyposis Syndrome, Hereditary Mixed, 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Why? PSYLIVED is a qualitative study that aims to understand the psychological experience of individuals living with inherited colorectal cancer. It addresses the question of how individuals cope emotionally and adapt to the unique challenges they face. This research sheds light on the emotional journey of those with inherited colorectal cancer, potentially leading to improved support services, interventions, and care practices tailored to their needs. The study seeks to enhance the well-being of patients undergoing genetic testing and contribute to better services and support practices.

What? PSYLIVED is a qualitative study that will employ reflexive Thematic Analysis methodology to explore the emotional responses and experiences of participants over time.

Who? The investigators are interested in interviewing between 30 to 66 individuals who have first-hand experience of being at risk or having an inherited colorectal cancer syndrome.

Where? While the study is conducted by the St Mark's Centre for Familial Intestinal Cancer, this study is open to individuals in the UK. Interviews will primarily be conducted via telephone or Microsoft Teams to facilitate accessibility. However, participants residing near London who prefer face-to-face interviews will be offered this option.

How? Each participant will take part in a one-hour audio-recorded interview where they will be asked to talk about their experiences. The interview will be recorded, so it can be transcribed word by word. During the transcription, the interview will be anonymised to ensure confidentiality. The responses will then be compared and analysed to create a result summary, along with interviews from other individuals with similar experiences. The study is set to commence in June 2024, with recruitment open for approximately two years.

DETAILED DESCRIPTION:
STUDY SUMMARY

Study Title: Opening Pandora's box: the Psychological Impacts of living with an inherited colorectal cancer predisposition syndrome Internal ref. no. (or short title): PSYLIVED Study Design: Qualitative Study Participants: Adults over 18 with an inherited predisposition or likelihood of inheriting colorectal cancer, offered genetic testing (with and without cancer history) Planned Size of Sample: 30-66 Follow up duration: After the initial interview, participants will not undergo any follow-up assessments. The screening questionnaire will determine the allocated study time-point for analysis. It's important to note that this study is not longitudinal.

Planned Study Period: 2024-2026 Research Question: What are the lived experiences and psychological adaptation processes of individuals diagnosed with inherited colorectal cancer over time?

PSYLIVED is a qualitative study exploring the psychological experience and long-term adaptation process of people living with inherited colorectal cancer. This project will recruit between 30 to 66 participants which will be allocated at one of the 3 time-points of the long-term adaptation process following the Family Systems Genetic Illness Model as articulated by Miller et al. in 2006 (1). The 3 time-points are:

1. Time-point 1: crisis I- pre-testing phase (before receiving genetic results)
2. Time-point 2: crisis II- post-testing phase (generally up 1 year post genetic testing. However, the team will follow a triage/evaluation system)
3. Time-point 3: long term adaptation phase (generally 1 year post genetic testing and beyond. However, the research team will use a triage/evaluation system) This approach will allow for a rich examination of how participants navigate the psychological impact of their genetic diagnosis across varying temporal contexts.

Each of the resulting six distinct datasets, as outlined in Table 1, will undergo individual analyses dedicated to uncovering the psychological adaptation processes at specific time-points. This methodological structure ensures a holistic exploration of the psychological trajectory experienced by individuals living with inherited colorectal cancer.

Furthermore, each analysis at distinct time-points will be refined by distinguishing between cancer and non-cancer patients. Subsequently, a synthesis of findings will be conducted through the comparison and combination of individual datasets. By generating a series of analytical sets, the study aims to provide a comprehensive understanding of the psychological journey undertaken by individuals living with inherited colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older, residing in the UK.
* Diagnosed with inherited colorectal cancer or likely to have inherited colorectal cancer and have been offered genetic testing for this reason.
* Possess the capacity to provide informed consent.
* Able to communicate in English.

Exclusion Criteria:

* Under 18 years old.
* Unable to communicate in English.
* Experience significant learning or communication difficulties.
* Reside outside of the UK.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 18 with an inherited predisposition or likelihood of inheriting colorectal cancer, offered genetic testing (with and without cancer history)
  This study population comprises individuals affected by the major inherited colorectal cancer syndromes, specifically focusing on Lynch syndrome and Polyposis syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
In-depth understanding of 'lived experiences' of people with or at risk of an inherited colorectal cancer Syndrome | 2 years.
  Detailed insights into the emotional responses, cognitive processes, and perceptions of individuals throughout their genetic diagnosis journey, providing a rich understanding of their lived experiences.
  This is a qualitative study using semi-structured interviews. Data from the qualitative semi-structured interviews will be used to address this outcome. Please note that no score or scale will be used in this research.

SECONDARY OUTCOMES:
Insight into psychological adaptation | 2 years
  understanding of how individuals psychologically adapt to the genetic diagnosis over time, identifying patterns of coping, emotional adjustments, and strategies employed to manage the psychological impact.
  This is a qualitative study using semi-structured interviews. Data from the qualitative semi-structured interviews will be used to address this outcome. Please note that no score or scale will be used in this research.
Contribution to patient wellbeing | 2 years
  Knowledge that contributes to improved patient care, by identifying psychological stressors, adaptive approaches, and potential areas for intervention, ultimately improving the overall well-being of individuals and families affected by inherited colorectal cancer.
  This is a qualitative study using semi-structured interviews. Data from the qualitative semi-structured interviews will be used to address this outcome. Please note that no score or scale will be used in this research.

CONTACTS AND LOCATIONS:
Locations (1):
- The St Mark's Centre for Familial Intestinal Cancer, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided